CLINICAL TRIAL: NCT05773482
Title: Effects of Breathing and Attention Training (BAT) on Pain Modulation in Healthy Individuals and Patients With Chronic Musculoskeletal Pain
Brief Title: Effects of Breathing and Attention Training (BAT) on Pain Modulation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: IRB202300172
Record Dates: First submitted 2023-03-06; First posted 2023-03-17 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-06

CONDITIONS: Fibromyalgia
MeSH Terms: conditions — Fibromyalgia | interventions — Respiration

STUDY DESIGN:
Intervention Model Description: This parallel study will be age & sex matched, and randomized.
Who Masked: Participant
Masking Description: Participants who do not receive BAT will be asked to perform deep breathing without mindfulness.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Breathing and Attention Training (BAT) (Experimental): Participants will be asked to do 20-minutes of focused breathing and attention training, involving focusing on taking deep breaths and becoming aware of the changing body sensations associated with breathing (mindfulness).
  Interventions: Behavioral: Breathing and Attention Training (BAT)
- Controlled Deep Breathing (Active Comparator): Participants will be asked to do 20-minutes of deep breathing and letting the body relax.
  Interventions: Behavioral: Breathing Control

INTERVENTIONS:
Behavioral: Breathing and Attention Training (BAT) — BAT is an instructor guided breathing technique over 20 min that will be applied once in a training session and approximately one week later in a testing session.
  Arms: Breathing and Attention Training (BAT)
Behavioral: Breathing Control — Controlled Breathing (without mindfulness) is an instructor guided breathing technique over 20 min that will be applied once in a training session and approximately one week later in a testing session.
  Arms: Controlled Deep Breathing

SUMMARY:
The hypersensitivity of fibromyalgia is associated with abnormal pain modulation within the CNS, but not with peripheral or central sensitization. Many brain areas that contribute to modulation of pain are known, but their testing is complex and expensive. Quantitative sensory testing is easier to perform and repeatable. Therefore, it will be used to evaluate the effects of Breathing Attention Training (BAT) on the hypersensitivity of FM participants. BAT is a form of mindfulness meditation shown to decrease FM symptoms and possibly pain sensitivity. We hypothesize that pain modulation of chronic pain patients is improved by BAT.

ELIGIBILITY:
Inclusion Criteria:

* Individuals diagnosed with fibromyalgia will have pain of duration > 6 months and meeting the 1990 Research Diagnostic Criteria for FM (ACR)
* Healthy, pain-free age matched controls without chronic pain

Exclusion Criteria:

* Personal or family history of photosensitive epilepsy
* Prior history of cancer or diabetes
* Patients must be willing to discontinue their analgesics, hypnotics, anxiolytics, or anti-depressants during the study period for at least 5 half-lives.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-04-03 (Actual); Primary Completion 2027-03-09 (Estimated); Study Completion 2028-03-09 (Estimated)

PRIMARY OUTCOMES:
Ratings of Painful and Painless Sensory Stimuli | 2 hr
  Ratings of painful and non-painful stimuli in FM subjects and HC will be obtained before and after BAT or Deep Breathing. Painful stimuli will include pressure stimuli. Painless stimuli will consist of flashing light stimuli.

CONTACTS AND LOCATIONS:
Overall Officials: Roland Staud, MD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No